CLINICAL TRIAL: NCT06386835
Title: Collagen Paste Injection Compared With Mucosal Advancement Flap for the Treatment of Fistula-in-ano: Single Centre Non-inferiority Randomised Controlled Trial
Brief Title: Collagen Paste vs Mucosal Advancement Flap for FIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kaori Futaba, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREC2021.724-T
Record Dates: First submitted 2024-04-22; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Fistula-in-ano
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen Paste (Experimental): Seton is removed, the fistula tract is de-epithelialised and collagen paste applied.
  Interventions: Procedure: Collagen Paste
- Mucosal Advancement Flap (Active Comparator): The internal opening is excised and is covered with a "U-shape" rectal mucosal flap
  Interventions: Procedure: Mucosal advancement

INTERVENTIONS:
Procedure: Collagen Paste — Collagen paste injection
  Arms: Collagen Paste
Procedure: Mucosal advancement — Mucosal advancement flap
  Arms: Mucosal Advancement Flap

SUMMARY:
The treatment for fistula-in-ano (FIA) remains a challenge to General and Colorectal Surgeons Worldwide. A variety of surgical treatments have been described for high anal fistulas, but none offers the panacea of fistula eradication with guaranteed preservation of continence. This study compares Collagen paste injection to mucosal advancement flap for the treatment of fistula-in-ano.

DETAILED DESCRIPTION:
Rectal advancement flaps have been advocated as a means of closing high fistulas with preservation of the external sphincter muscle. With this technique, it shows promising results with success rate of approximately 60%. However, complications have been reported, in particular with a change of continence in 30-35% of patients.

Collagen paste is a novel sphincter-preserving method for fistula closure. Permacol (Medtronic, USA) is a sterile acellular cross-linked porcine dermal collagen matrix suspension. The paste-like suspension form a matrix that accelerates neovascularization, cellular infiltration which promotes healing and fistula closure. The theoretical benefits of paste form compared to previous collagen plug design is that the collagen can moulded into the fistula cavity or tract. This allows better tissue contact with the collagen thus improves healing and reduces the chance of dislodgement. Limited data is available to date. Success rates of collagen paste range from 47.6% to 63%. Hence it has a potential to be the first-line treatment for high FIA with low complication rates and without causing disruption to the anal sphincter complex.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of high cryptoglandular fistula-in-ano.
* Patients must have undergone a prior EUA to characterise the nature of the fistula.
* The fistula tract should be ≥ 2 cm in length.
* Only a single internal fistula opening should be present at EUA, such that the fistula is suitable for treatment by insertion of a seton drain.
* Patients must have been treated with a draining seton for a minimum period of 6 weeks prior to randomisation.
* Patients must be aged ≥ 18 years and able to provide informed consent.
* Fistulas must be of cryptoglandular aetiology.

Exclusion Criteria:

* Unable/unwilling to provide informed consent.
* Contraindication to general anaesthesia or spinal anaesthesia.
* Low trans-sphincteric fistulas.
* Non-cryptoglandular fistulas (e.g. Crohn's disease, obstetric, irradiation, malignant, etc.).
* Other perineal fistulas (e.g. rectovaginal fistulas, pouch-vaginal fistulas, etc.).
* Complex disease in which more than one internal fistula opening is present and requiring concurrent insertion of more than one fistula plug.
* Clinical evidence of active perianal sepsis. In the event that there is disagreement between clinical and radiological assessment of active sepsis/collection, the clinical opinion will prevail.
* Cultural or religious objection to the use of pig tissue.
* Absolute contraindication to magnetic resonance imaging (MRI) (e.g. cardiac pacemaker).
* Patients with recurrent anal fistulas previously treated with a fistula plug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical healing of Fistula-in-ano | 1 year
  Clinical healing of the fistula-in-ano

SECONDARY OUTCOMES:
30-day morbidity | 30 days
  30-day morbidity using Clavien-Dindo classification
Quality of life score | 1 year
  Assess effect on Quality of life post operatively using Short Form 36 Health Survey
Postoperative pain score | 1 week
  assessment of postoperative pain using visual analog score from 0 (no pain) to 10 (severe pain)
Faecal incontinence rate | 1 year
  Assess postoperative effect on continence
Hospital readmission rate | 1 year
  Assess hospital re-admission rate

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Department of Surgery, Chinese University of Hong Kong, Shatin, New Territories
  - Prince of Wlaes Hospital, Shatin